CLINICAL TRIAL: NCT02028247
Title: 2/3 Treatment of Anxiety in Autism Spectrum Disorder
Brief Title: Psychotherapy for Anxiety in Children With Autism Spectrum Disorder
Acronym: TAASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Temple University (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Eric Storch, McIngvale Presidential Endowed Chair & Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NICHD CBT for ASD; NCT02111395 (obsolete NCT alias)
Record Dates: First submitted 2014-01-02; First posted 2014-01-07 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Autism Spectrum Disorders; Autism; Asperger's Syndrome; Pervasive Developmental Disability - Not Otherwise Specified; Obsessive-compulsive Disorder; Social Phobia; Generalized Anxiety Disorder; Specific Phobia; Separation Anxiety Disorder
Keywords: Autism spectrum disorders; Autism; Asperger's syndrome; Pervasive developmental disability - not otherwise specified; obsessive-compulsive disorder; Social phobia; Generalized anxiety disorder; Specific phobia; Separation anxiety disorder; Counseling; Cognitive-behavioral therapy; Psychotherapy
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Asperger Syndrome; Obsessive-Compulsive Disorder; Phobia, Social; Generalized Anxiety Disorder; Phobia, Specific; Anxiety, Separation | interventions — Behavior Therapy; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Personalized Cognitive-behavioral therapy (Experimental): Personalized Cognitive-behavioral therapy involves 16 weekly individual therapy sessions, up to 90 minutes each, based on a treatment protocol that has been designed specifically for youth with high-functioning autism spectrum disorders.
  Interventions: Behavioral: Personalized Cognitive-behavioral therapy
- Standard Practice Cognitive-behavioral therapy (Active Comparator): Standard Practice Cognitive-behavioral therapy involves 16 weekly individual therapy sessions, up to 60 minutes each, based on a treatment protocol that represent the standard practice psychotherapy for anxiety that has been found to be effective in multiple trials in youngsters without autism spectrum disorders.
  Interventions: Behavioral: Standard Practice Cognitive-behavioral therapy
- Treatment as Usual (Other): Participants randomized to the TAU condition will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions) for a 16-week period. Treatment changes (e.g., medication increase, starting psychotherapy in community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Personalized Cognitive-behavioral therapy
  Other Names: Behavioral Interventions for Anxiety in Children with Autism
  Arms: Personalized Cognitive-behavioral therapy
Behavioral: Standard Practice Cognitive-behavioral therapy
  Other Names: Coping Cat
  Arms: Standard Practice Cognitive-behavioral therapy
Behavioral: Treatment as Usual
  Arms: Treatment as Usual

SUMMARY:
Anxiety disorders affect 40 to 50% of children with autism spectrum disorders (ASD), contributing to substantial distress and impairment. The goal of this study is to examine the effectiveness of a personalized type of psychotherapy against standard-care psychotherapy for addressing anxiety in youth with ASD.

DETAILED DESCRIPTION:
Autism spectrum disorders (ASD) are common neurodevelopmental syndromes affecting 1% of U.S. children. Comorbid anxiety disorders affect 40 to 50% of children with ASD, causing substantial distress and impairment over and above that caused by ASD alone. Although standard practice cognitive-behavioral therapy (CBT) has been established as an efficacious and safe treatment for anxiety disorders among typically developing youth, its utility in comorbid cases with ASD remains unknown. To date, no studies have experimentally compared standard practice CBT to a cognitive-behavioral intervention that has been personalized for children with a comorbid presentation of anxiety and ASD. Accordingly, we are proposing a randomized controlled trial to be conducted at three treatment sites to evaluate the efficacy of personalized CBT for anxiety in ASD (Behavioral Intervention for Anxiety in Children with Autism: BIACA) relative to standard practice CBT for anxiety (Coping Cat program). Furthermore, this study will employ a waitlist control group to assess the efficacy of each CBT arm relative to the absence of treatment (i.e., a Waitlist control arm). The proposed research will: (1) examine the efficacy of BIACA relative to Coping Cat, which represents standard practice treatment, and the efficacy of both these treatments relative to a waitlist control group, (2) evaluate the maintenance of treatment gains, (3) examine the impact of personalized intervention on functional outcomes. A total of 201youth across 3 study locations (ages 8-13 years) with ASD and co-occurring anxiety will be randomly assigned to one of the three conditions. The three recruitment sites for this study are University of California, Los Angeles, the University of South Florida (USF), and Temple University. Considering the rising number of children diagnosed with ASD together with the frequency and severity of comorbid anxiety, the proposed work is tailored to the unique needs of youth with ASD and will provide a timely contribution to public health efforts.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient boys and girls with ASD between the ages 7-13 years at consent/assent.
* The child meets criteria for ASD.
* The child meets criteria for clinically significant anxiety symptoms.
* The child has a Full Scale and Verbal Comprehension Intelligence Quotient >70 as assessed on the Wechsler Intelligence Scale for Children-IV or another acceptable Intelligence Quotient test.

Exclusion Criteria:

* Receiving concurrent therapy targeting anxiety, social skills training with homework, or behavioral interventions (e.g., applied behavior analysis). This excludes academic tutoring, occupational therapy, speech therapy, school counseling that is no more than 60 minutes per week in duration, school aides, and social skills training groups that do not include homework and are no more than 60 minutes/week in duration.
* (a) Current clinically significant suicidality or (b) individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
* Child has been nonresponsive to an adequate trial of CBT for anxiety within the previous 2 years.
* Lifetime bipolar disorder, schizophrenia or schizoaffective disorder.
* Initiation of an antidepressant medication within 12 weeks before study enrollment or an antipsychotic medication 6 weeks before study enrollment or the child has changed the dose of an established medication within 8 weeks before study enrollment (4 weeks for antipsychotic) or during psychotherapy (unless the dose is lowered because of side effects).

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Storch, Ph.D., Principal Investigator — University of South Florida; Jeff Wood, Ph.D., Principal Investigator — University of California, Los Angeles; Philip C Kendall, Ph.D., Principal Investigator — Temple University
Locations (1):
- Rothman Center for Neuropsychiatry, University of South Florida, St. Petersburg, Florida, United States

REFERENCES:
- [Derived] Wood JJ, Rosenau KA, Muscatello V, Cooper K, Wood KS, Kendall PC, Storch EA. Cognitive Behavioral Therapy for Autistic School-Aged Children with Interfering Anxiety: Impact on Caregiver-Defined Goals. J Autism Dev Disord. 2025 May 8. doi: 10.1007/s10803-025-06852-6. Online ahead of print. PMID 40338510
- [Derived] Storch EA, Wood JJ, Guzick AG, Small BJ, Kerns CM, Ordaz DL, Schneider SC, Kendall PC. Moderators of Response to Personalized and Standard Care Cognitive-Behavioral Therapy for Youth with Autism Spectrum Disorder and Comorbid Anxiety. J Autism Dev Disord. 2022 Feb;52(2):950-958. doi: 10.1007/s10803-021-05000-0. Epub 2021 Apr 7. PMID 33826038
- [Derived] Wood JJ, Kendall PC, Wood KS, Kerns CM, Seltzer M, Small BJ, Lewin AB, Storch EA. Cognitive Behavioral Treatments for Anxiety in Children With Autism Spectrum Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2020 May 1;77(5):474-483. doi: 10.1001/jamapsychiatry.2019.4160. PMID 31755906

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two-hundred and fourteen children between 7-13 years (M=9.96, SD=1.76) were recruited through referrals, advertisements, and the patient flow of three university-based mental health clinics. Recruitment began April 2014 and final data were collected around January 2017.
Pre-assignment Details: Of the 214 participants enrolled in the study, a total of 47 children were excluded before assignment to groups because they did not meet eligibility criteria (did not meet IQ criteria (n=6); did not meet anxiety criteria or anxiety was not primary (n=16); no autism spectrum disorder criteria (n=17); parent unwilling or unable to adhere to study procedures (n=7); child needed a higher level of care (n=1)). Thus, only 167 children were assigned across the three groups.
Groups:
- Personalized Cognitive-behavioral Therapy: Personalized Cognitive-behavioral therapy involves 16 weekly individual therapy sessions, up to 90 minutes each, based on a treatment protocol that has been designed specifically for youth with high-functioning autism spectrum disorders.
  Personalized Cognitive-behavioral therapy
- Standard Practice Cognitive-behavioral Therapy: Standard Practice Cognitive-behavioral therapy involves 16 weekly individual therapy sessions, up to 60 minutes each, based on a treatment protocol that represent the standard practice psychotherapy for anxiety that has been found to be effective in multiple trials in youngsters without autism spectrum disorders.
  Standard Practice Cognitive-behavioral therapy
- Treatment as Usual: Participants randomized to the TAU condition will be instructed to continue receiving their prior interventions as recommended by their providers (e.g., psychotherapy, social skills training, behavioral interventions, family participation in family therapy or a parenting class, or pharmacological interventions) for a 16-week period. Treatment changes (e.g., medication increase, starting psychotherapy in community) are not prohibited and will be monitored. Thus, treatment will continue as it would in standard practice; and will be monitored through periodic study assessment.
  Treatment as Usual
Period: Overall Study
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
Started | 77 | 71 | 19
Completed | 67 | 59 | 15
Not Completed | 10 | 12 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual | Total
Number analyzed (Participants) | 77 | 71 | 19 | 167
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 77 | 71 | 19 | 167
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.71 (1.86) | 10.03 (1.66) | 10.05 (1.75) | 9.90 (1.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 12 | 0 | 33
  Male | 56 | 59 | 19 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 3
  Asian | 6 | 3 | 1 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 2 | 3 | 11
  White | 58 | 57 | 13 | 128
  More than one race | 0 | 4 | 1 | 5
  Unknown or Not Reported | 5 | 4 | 1 | 10
Region of Enrollment [Number; unit: participants]
  United States | 77 | 71 | 19 | 167

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Anxiety Severity on the Pediatric Anxiety Rating Scale After 16 Weeks of Treatment.
Description: This measure is administered by a clinician and assesses anxiety symptom severity on a scale from 0-25 with higher scores corresponding to worse anxiety.
Time Frame: Baseline and After 16 Weeks of Treatment
Population: Not all participants who were randomized to each of the intervention arms completed the Pediatric Anxiety Rating Scale (at baseline and/or post-treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 77 | 69 | 19
units on a scale
  Baseline | 3.43 (0.48) | 3.47 (0.47) | 3.28 (0.39)
  Post-treatment: number analyzed (Participants) | 66 | 59 | 18
  Post-treatment | 2.13 (0.91) | 2.43 (0.70) | 2.93 (0.59)

2. Secondary Outcome: Percentage of Participants With Positive Treatment Response as Assessed by the Clinical Global Impressions-Improvement Scale
Description: The Clinical Global Impressions-Improvement scale (CGI-I) was completed by a clinician after 16 weeks of treatment. The CGI-I assesses the severity of anxiety on a 7 point scale, ranging from 1 (very much improved) to 7 (very much worse). A rating of 1 or 2 on the CGI-I designated a positive treatment response.
Time Frame: After 16 weeks of treatment
Population: Of the 167 participants assigned to groups, only 145 completed treatment (67 in personalized CBT, 60 in standard CBT, and 18 in treatment as usual). For 3 participants (1 in personalized CBT and 2 in standard CBT), the Clinical Global Impressions-Improvement Scale was not completed at the end of treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 66 | 58 | 18
percentage of participants | 92.42 | 81.03 | 11.11

3. Secondary Outcome: Change From Baseline in Anxiety/Depression Severity on the Child Behavior Checklist After 16 Weeks of Treatment.
Description: The Child Behavior Checklist (CBCL) is completed by parents and the anxiety/depression subscale of the CBCL was used to assess anxiety/depression symptomatology. The CBCL anxiety/depression subscale is rated on a 3-point scale, ranging from 0 (Not true) to 2 (Very True), with higher scores indicating more symptoms.
Time Frame: Baseline and After 16 weeks of treatment
Population: Not all participants who were randomized to each of the intervention arms completed the Child Behavior Checklist (at baseline and/or post-treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 76 | 69 | 17
units on a scale
  Baseline | 0.83 (0.39) | 0.88 (0.39) | 0.73 (0.28)
  Post-treatment: number analyzed (Participants) | 63 | 55 | 17
  Post-treatment | 0.51 (0.29) | 0.69 (0.34) | 0.77 (0.27)

4. Secondary Outcome: Change From Baseline in Anxiety Related Impairment as Measured by the Childhood Anxiety Impact Scale After 16 Weeks of Treatment.
Description: The Childhood Anxiety Impact Scale (CAIS) is a questionnaire completed by parents about the impact of the child's anxiety on functioning in three situational categories (i.e., school, social, and family functioning). The CAIS is rated on a 4-point scale, ranging from 0 (not at all) to 3 (very much). The CAIS items are summed and sorted into 3 subscales, corresponding to each situational category: school, social, and family. For all 3 subscales, higher scores correspond to more associated impact in that area.
Time Frame: Baseline and After 16 weeks of treatment
Population: Not all participants who were randomized to each of the intervention arms completed the Childhood Anxiety Impact Scale (at baseline and/or post-treatment).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
Number analyzed (Participants) | 76 | 70 | 18
units on a scale
  Baseline - CAIS School: number analyzed (Participants) | 76 | 69 | 18
  Baseline - CAIS School | 1.38 (0.61) | 1.48 (0.60) | 1.19 (0.70)
  Post - CAIS School: number analyzed (Participants) | 63 | 54 | 17
  Post - CAIS School | 0.77 (0.57) | 0.88 (0.54) | 1.24 (0.51)
  Baseline - CAIS Social: number analyzed (Participants) | 76 | 70 | 17
  Baseline - CAIS Social | 0.97 (0.56) | 0.96 (0.62) | 0.70 (0.54)
  Post - CAIS Social: number analyzed (Participants) | 64 | 55 | 17
  Post - CAIS Social | 0.49 (0.42) | 0.65 (0.54) | 0.80 (0.50)
  Baseline - CAIS Family: number analyzed (Participants) | 75 | 70 | 18
  Baseline - CAIS Family | 1.16 (0.63) | 1.12 (0.62) | 0.98 (0.44)
  Post - CAIS Family: number analyzed (Participants) | 64 | 55 | 17
  Post - CAIS Family | 0.65 (0.49) | 0.73 (0.51) | 0.88 (0.60)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: During the course of the acute intervention (16 week duration).
Arm/Group | Personalized Cognitive-behavioral Therapy | Standard Practice Cognitive-behavioral Therapy | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/77 | 0/71 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/71 | 0/19
Other Adverse Events (participants affected / at risk) | 0/77 | 0/71 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-04): https://cdn.clinicaltrials.gov/large-docs/47/NCT02028247/Prot_SAP_000.pdf